CLINICAL TRIAL: NCT02399605
Title: Subcutaneous Electrical Stimulation in the Prevention of Postoperative Ileus in Colorectal Surgery
Brief Title: Subcutaneous Electrical Stimulation in the Prevention of Postoperative Ileus
Acronym: SESPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Pedro Moya, PhD, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Cirugia1
Record Dates: First submitted 2015-03-10; First posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Ileus
MeSH Terms: conditions — Ileus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No intervention, group control.
- Stimulation (Experimental): Subcutaneous Electrical Intervention
  Interventions: Other: Stimulation

INTERVENTIONS:
Other: Stimulation — Subcutaneous abdominal electrical stimulation
  Arms: Stimulation

SUMMARY:
Assess whether the application of electrical stimulation in patients undergoing subcutaneous colon cancer in a Multimodal Rehabilitation Program (Fast track) decreases the incidence of postoperative ileus, improving the results of morbidity and mortality, hospitalization and health care costs.

DETAILED DESCRIPTION:
Prospective randomized study on the application of subcutaneous abdominal electrical stimulation in the postoperative of colonic surgery and its relationship with the appearance of postoperative ileus.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colorectal surgery.
* Signing informed consent.

Exclusion Criteria:

* Patients with no oral nutrition (dysphagia, esophageal stricture, pyloric stenosis)
* Patients with contraindications for electrical stimulation.
* Psychiatric Disorders
* HIV
* Pregnant or breastfeeding
* intestinal obstruction
* uncontrolled infection
* ASA IV
* No acceptance or failure to follow protocol multimodal rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Time to first flatus | Participants will be followed for the duration of hospital stay, an expected average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Moya, PhD, Principal Investigator — HGU ELCHE
Locations (2):
- Spain (2):
  - Pedro Moya, Elche, Spain
  - Pedro Moya, Alicante